CLINICAL TRIAL: NCT01558050
Title: The Effect of a Commercially Available Red Rice Nutrition Supplement on Serum Lipids
Brief Title: the Effect of a Red Rice Nutrition Supplement on Cholesterol Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Veronique Verhoeven, professor dr, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RR001
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Cholesterol Level; HDL Level; LDL Level; TG Level
MeSH Terms: interventions — red yeast rice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- red rice (Experimental): commercially available red rice nutritionial supplement
  Interventions: Dietary Supplement: red rice supplement
- placebo (Placebo Comparator): placebo capsules
  Interventions: Dietary Supplement: red rice supplement

INTERVENTIONS:
Dietary Supplement: red rice supplement — patricipants take a red rice supplement or placebo daily for 8 weeks

SUMMARY:
In this study the investigators investigate the effect of a red rice product on plasma lipids in a sample of physicians and/or their family members.

After a baseline measurement of cholesterol, HDL, LDL and TG, participants are randomised to receive a commercially available red rice product or placebo. After a period of 8 weeks, lipid levels are measured again.

ELIGIBILITY:
Inclusion Criteria:

* total fasting cholesterol > 200mg/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
fasting cholesterol, LDL, HDL, TG level | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp, Wilrijk, Belgium

REFERENCES:
- [Derived] Verhoeven V, Lopez Hartmann M, Remmen R, Wens J, Apers S, Van Royen P. Red yeast rice lowers cholesterol in physicians - a double blind, placebo controlled randomized trial. BMC Complement Altern Med. 2013 Jul 18;13:178. doi: 10.1186/1472-6882-13-178. PMID 23866314